CLINICAL TRIAL: NCT03477266
Title: Effectiveness of Mouth Dissolving Mosapride Tablets on Enhancing Gut Recovery After Cesarean Section: Randomized Double-blind, Placebo-controlled Clinical Trial
Brief Title: Mouth Dissolving Mosapride Tables Enhance Post Cesarean Gut Recovery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, ashraf nassif mahmoud elmantwe,MD, Assistant professor, Benha University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Ashrafnassif2002@yahoo.com
Record Dates: First submitted 2018-02-21; First posted 2018-03-26 (Actual); Last update posted 2018-08-14 (Actual); Status verified 2018-08

CONDITIONS: Prevention of Postoperative Ileus
Keywords: Postoperative ileus; mosapride; mouth dissolving tablets; Intraoperative vomiting
MeSH Terms: interventions — mosapride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Color coded active tablets backed in red while identical dummy tablets coded in blue,both tablets are physically identical and usually no anticipated noticed side effects from mosapride
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mouth dissolving mosapride (Experimental): Fluxopride 5mg of Macryrl egypt 2 tablets one day before and immediately after elective cesarean section every 8hour for maximum of 5 days
  Interventions: Drug: Mosapride
- Placebo mouth dissolving tablets (Placebo Comparator): Dummy identical tablets taken in the same way
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Mosapride — Intake mouthly dissolving mosapride tablets in immediate post cesarean section
  Other Names: Fluxopride
  Arms: Mouth dissolving mosapride
Drug: Placebo Oral Tablet — Dummy identical tablets to mouthly dissolving mosapride tablets
  Other Names: Placebo
  Arms: Placebo mouth dissolving tablets

SUMMARY:
Giving women one day before and immediately after cesarean section a mouthly dissolving mosapride tablets 2every every 8 hours for maximum of 5 days ,or getting recovered gastrointestinal functions And assess preoperative gastrointestinal functions

DETAILED DESCRIPTION:
Uncomplicated post cesarean women one day before and immediately after elective cesarean receive 2 mouthly dissolving mosapride tablets every 8 hours maximum for 5 days and clinical care giver follow the woman's gastrointestinal functions, including intraoperative and postoperative nausea vomiting, passing flatus, hearing intestinal sounds, passing stools, occurring of paralytic ileus, length of the hospital stay

ELIGIBILITY:
Inclusion Criteria:

* all women undergoing elective cesarean section

Exclusion Criteria:

* prior abdominal surgery, abdominal adhesion, chronic constipation, allergy to mosapride

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — After cesarean section
Enrollment: 400 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2018-08-01 (Actual)

PRIMARY OUTCOMES:
Time of first flatus | 96 hours postoperative
  Clinical

SECONDARY OUTCOMES:
Paralytic ileus incidence and its severity | 7days
  Clinical
Toleration of fluids and solids intake | 2 weeks postoperative
  Clinical
Incidence of intraoperative and postoperative nausea and vomiting | Intraoperative and 2 weeks postoperative
  Clinical
First defecation | 2 weeks postoperative
  Clinical

CONTACTS AND LOCATIONS:
Overall Officials: Ashraf N Elmantwe, MD, Principal Investigator — Benha University
Locations (1):
- Ashraf nassif Elmantwe, Banhā, Elqalopia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Once data collected and analyzed and published
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: When data became available and for ever
Access Criteria: Any